CLINICAL TRIAL: NCT03555747
Title: Molecular Analysis of Gingival Crevicular Fluid in Response to the Magnitude of Orthodontic Force: a Longitudinal Randomized Split-mouth Study
Brief Title: Gingival Crevicular Fluid Cytokine Levels in Response to Orthodontic Forces
Acronym: GCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Collaborators: Ege University (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Beral Afacan, Assistant Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: bafacan09
Record Dates: First submitted 2018-05-19; First posted 2018-06-13 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Orthodontic Tooth Movement
Keywords: Canine distalization; Gingival crevicular fluid; Cytokines; Orthodontic force; Periodontium; Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Canine distalization by 75 g force (Other): Canine was distalized using a continuous force of 75 g with nickel-titanium closed coil springs.
  Interventions: Other: Canine distalization
- Canine distalization by 150 g force (Other): Canine was distalized using a continuous force of 150 g with nickel-titanium closed coil springs.
  Interventions: Other: Canine distalization

INTERVENTIONS:
Other: Canine distalization — GCF was sampled from the mesial (tension) and distal (pressure) sides of maxillary right and left canines immediately before appliance placement (baseline) and after force application (24 hours and 28 days)
  Other Names: Gingival crevicular fluid collection

SUMMARY:
The aim of this randomized split-mouth study was to quantify simultaneously 30 analytes including cytokines, chemokines and growth factors in gingival crevicular fluid (GCF) in response to different magnitudes of forces during maxillary canine distalization. The upper right and left canines were distalized using a continuous force of 75 g or 150 g in 15 individuals who had Class II division I malocclusion requiring bilateral extraction of maxillary first premolars. GCF samples were obtained from the tension and the pressure side of each canine at appliance placement and after force application at 24 hours and 28 days. A multiplexed bead immunoassay was used to quantify 30 analytes simultaneously. The effect of force, side and time on the analyte levels were analyzed with Brunner-Langer method.

DETAILED DESCRIPTION:
Patient selection:

Fifteen orthodontic patients with class II division I malocclusion, who required the extractions of maxillary first premolars bilaterally, distal canine movement, and maximum anchorage control as a part of fixed orthodontic treatment plan were invited to participate in the study. All subjects were in good general health with clinically and radiological healthy periodontal tissues (the probing depths ≤3 mm, full-mouth plaque and bleeding score ≤15%, and no bone loss radiographically). Patients were excluded if they were smokers, had had previous orthodontic treatment, had taken a course of anti-inflammatory drugs within 1 month and antimicrobial agents in the previous 3 months prior to the start of the study.

Experimental Design:

The first premolars were extracted at least 20 days prior to the distalization of the canines. Ten days prior to the application of orthodontic force all subjects underwent full-mouth scaling and oral hygiene instructions to ensure optimal plaque control and oral hygiene instruction was reinforced throughout the whole study period. In each patient, two mini-screw implants (1.5 mm in diameter and 8.0 mm in length) were placed bilaterally into the inter-radicular bone between the maxillary second premolar and first molar in the attached gingiva.The upper right and left canines of the same patient were randomly distalized using a continuous force of 75 or 150 g with nickel-titanium closed coil springs. Simple randomization by flipping a coin was used to determine the assignment of each site for two different forces.

GCF sampling:

GCF was sampled from the mesial (tension) and distal (pressure) sides of maxillary right and left canines immediately before appliance placement (baseline) and after force application at 24 hours and 28 days without any reactivation of the coil spring. Baseline measurements of maxillary canines served as a control.

Clinical Periodontal Measurements:

Periodontal clinical parameters including probing depth, clinical attachment loss, gingival index and plaque index were recorded at mesial and distal sites of distally moved canines at baseline and 24 hours and 28 days after force application. All clinical periodontal examinations were performed by a single calibrated periodontist who blinded to the groups using a manual periodontal probe.

Multiplex assay& Quantification of inflammatory mediators:

A commercially available multiplex panel including thirty proteins was used to evaluate GCF content on the Luminex®200 platform.

Determination of the amount of tooth movement:

The distance of maxillary canine movement was measured from the cusp tip of a distally moved canine to the buccal groove of the first permanent molar by using a digital caliper with a sensitivity of ±0.01 mm.

Statistical Analysis:

The data was analysed using a statistical software package. The effect of force, side and time on the analyte levels were analyzed with Brunner-Langer method.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* Non-smoker
* Orthodontic patients with class II division I malocclusion

Exclusion Criteria:

* Orthodontic treatment history
* Use of anti-inflammatory drugs within one month
* Use of antibiotics within last three months

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2015-05-29 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Gingival crevicular fluid protein content change | Change from baseline to 24 hours and to 28 days after force application
  pg/ml

SECONDARY OUTCOMES:
Probing pocket depth change | Change from baseline to 24 hours and to 28 days after force application
  mm
Clinical attachment level change | Change from baseline to 24 hours and to 28 days after force application
  mm
The amount of tooth movement | Change from baseline to 28 days after force application
  mm

REFERENCES:
- [Derived] Afacan B, Ozturk VO, Gecgelen Cesur M, Kose T, Bostanci N. Effect of orthodontic force magnitude on cytokine networks in gingival crevicular fluid: a longitudinal randomized split-mouth study. Eur J Orthod. 2019 Mar 29;41(2):214-222. doi: 10.1093/ejo/cjy068. PMID 30321318